CLINICAL TRIAL: NCT04374838
Title: Effect of COVID-19 Pandemic on Pediatric Cancer Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Mahmoud Motaz Elzembely, Lecturer of Pediatric Oncology, South Egypt Cancer Institute
Other Study IDs: COVID-19 and Pediatric Cancer
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: Pediatric Oncology, COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational cohort study to assess the effects of COVID19 on pediatric cancer care in Egypt and the Arab World through a survey applied to pediatric oncologists who will be interviewed either directly or through the internet to assess the effect of COVID 19 on pediatric cancer care

DETAILED DESCRIPTION:
Corona viruses are single stranded enveloped RNA viruses with helical capsids. They infect wide variety of hosts including humans and animals. Coronavirus disease 2019 (COVID-19) was first described in December 2019 in Wuhan, the capital of China's Hubei province. A novel corona virus named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was identified as the causative organism. On 30 Jan 2020, WHO declared COVID-19 as a Public Health Emergency of International Concern (PHEIC). Subsequently on 11 March 2020, WHO declared COVID-19 as a pandemic. On April 30, 2020; 3,239,220 confirmed cases were diagnosed across the globe with 228,860 deaths. The united states has the highest number of cases followed by spain and Italy. The first confirmed case of COVID-19 in Egypt was reported on 14 February 2020. As of April 30, 2020, there have been 5,537 confirmed cases, 1381 recovered and 392 deaths The overall global incidence of cancers in children aged 0-14 years is 140·6 per million, whereas, It's 130.9 per million in Egypt. Although cancer is a rare disease among children and adolescent, It's one of the leading causes of death. The prognosis of childhood cancer has significantly improved over the past decades with 5-year survival rates improved from 58% in the mid-1970 to around 83% in 2008-2014.

Little is known about the effects of COVID-19 on children with cancer. Children with cancer face numerous challenges during COVID-19 pandemic. Children with cancer are immunocompromised because of cancer or anti-cancer therapy. They have to be hospitalized to receive their anti-cancer therapy. The major problem we-as pediatric oncologist- face nowadays is how to organize pediatric cancer care in the COVID-19 ERA.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric oncologists working in cancer centers in Egypt and the Arab world during COVID 19 pandemic

Exclusion Criteria:

* Pediatric oncologists not caring for patients during COVID 19 pandemic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric oncologists working in cancer centers in Egypt and the Arab world will be interviewed either directly or through the internet to assess the effect of COVID 19 on pediatric cancer care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
pediatric cancer care pattern during COVID 19 pandemic | 3 months
  Patterns of data will be mined to understand pediatric cancer care adaptation during COVID 19 pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Steliarova-Foucher E, Colombet M, Ries LAG, Moreno F, Dolya A, Bray F, Hesseling P, Shin HY, Stiller CA; IICC-3 contributors. International incidence of childhood cancer, 2001-10: a population-based registry study. Lancet Oncol. 2017 Jun;18(6):719-731. doi: 10.1016/S1470-2045(17)30186-9. Epub 2017 Apr 11. PMID 28410997